CLINICAL TRIAL: NCT04945278
Title: Study of Self-Recognition and Self/Other Distinction Disorders in Patients With Psychological Vulnerability (ALTER EGO)
Brief Title: Study of Self-Recognition and Self/Other Distinction Disorders in Patients With Psychological Vulnerability
Acronym: ALTER-EGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC20.0283
Record Dates: First submitted 2021-04-22; First posted 2021-06-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Psychosis of Childhood Borderline; Psychotic Disorder
Keywords: Mental Vulnerability; Self-recognition; Psychosis High-Risk State; Self-other Distinction; Double Mirror Paradigm; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Prospective interventional case / control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Both patients and healthy volunteers arms will undergo the double mirror test within a day.
  But the patients arm will additionally respond to the EASE test.
  Interventions: Other: Double mirror device ALTER-EGO; Other: EASE test
- Healthy volunteers (Other): Both patients and healthy volunteers arms will undergo the double mirror test within a day.
  Interventions: Other: Double mirror device ALTER-EGO

INTERVENTIONS:
Other: Double mirror device ALTER-EGO — The patient and his matched healthy volunteer will be placed on each side of the double mirror device ALTER-EGO. Both sides will be lightened alternatively or at the same time by lights, so according to the light intensity, the subject will see himself in a mirror or the other person throw a classic window. The light intensity will vary from 0 to 100% and to 100% to 0% alternatively from each side of the mirror. At each 10% variation of one side, both patient and volunteer will have to answer that question : "who do you see more : him/her or yourself ?"
Other: EASE test — The patient will have to answer the EASE test which is a specific test to detect patient with high risk of psychosis or schizophrenia
  Arms: Patients

SUMMARY:
The main objective of this study is to establish whether there are differences in self-recognition and self/other distinction in subjects with psychological vulnerability compared to healthy volunteer controls.

DETAILED DESCRIPTION:
This study is based on the properties of the double mirror "Alter Ego" which is a device that appears as a double-sided mirror surrounded by light diodes whose intensity can be varied. Thanks to this variation of luminosity, this special paradigm creates morphs between two real subjects seated on both sides, resulting in different faces, each morphed to a varying extent.

In this task, participants watch a double mirror in which a picture of their own face gradually transforms into the face of an unfamiliar other (self-to-other direction) or vice versa (other-to-self direction), and indicate at which point they judge the morph to look more like the target face than the starting face.

The comparison of the thresholds obtained by different individuals makes it possible to establish whether there could be differences between subjects with psychological vulnerability and healthy controls and to explore hypothetical links between self/other distinction abilities and symptoms of psychological vulnerability .

ELIGIBILITY:
Inclusion criteria for patients:

* Aged from 15 to 25 years
* Subject meeting the Ultra High Risk criteria at CAARMS and / or SPI-A
* Signature of the consent (participants and parents for minors)
* Subject affiliated to the social security scheme or benefiting from such a scheme

Inclusion criteria for healthy volunteers:

* Aged from 15 to 25 years
* Subject not familiar to the patient to whom it is matched
* Signature of the consent (participants and parents for minors)
* Subject affiliated to the social security scheme or benefiting from such a scheme

Exclusion Criteria for both patients and healthy volunteers:

* History of epilepsy and / or migraine (due to the epileptogenic potential of light stimuli)
* Refusal of participation of the minor even if the legal representatives want the subject to participate in the study
* Claustrophobia
* Wearing glasses
* Abnormal right and left visual acuity without contact lenses
* Distinctive signs on the face which cannot be temporarily removed
* Subject under legal protection (curators / guardianship) or deprived of liberty

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Average of the three M1 | Inclusion
  Average of the three M1 thresholds obtained from the "round trip" manipulation repeated three times, the M1 threshold corresponding to the level of luminosity from which a subject begins to recognize himself when his own image gradually appears (during the passage of the condition glass in mirror condition).

SECONDARY OUTCOMES:
The average of the three M2 | Inclusion
  The average of the three M2 thresholds obtained from the "round trip" manipulation repeated three times, the M2 threshold corresponding to the level of brightness from which a subject ceases to recognize himself to recognize the other (passage of the mirror mode to window mode).
Results to tests for early prodromal symptoms assessed by SPI-A (Schizophrenia Prediction Instrument for Adults) | Inclusion
  • Hetero-questionnaire of SPI-A : intensity, type and frequency of symptoms : The answer "yes" to the COPER (Cognitive-Perceptive Basic Symptoms) and / or COGDIS (Cognitive Disturbances) criteria points to at risk mental state.
Results to tests for early prodromal symptoms assessed by PQ16 (Prodromal Questionnaire - 16) | Inclusion
  • Self-administered questionnaire PQ16 : intensity, type and frequency of symptoms : The minimum score is 0 and maximum 16 meaning a higher state of risk.
Results to tests for early prodromal symptoms assessed by EASE(xamination of Anomalous Self-Experience) | Inclusion
  • Self-experience anomalies evaluation scale : EASE, Parnas, 2003), until now not carried out as part of the routine monitoring of CEVUP (Consultation d'Evaluation de la VUlnérabilité Psychique = Psychic Vulnerability Assessment Consultation) patients : score between 0 and 57, the higher the score, the greater the risk of psychosis
Results to tests for later prodromal symptoms | Inclusion
  CAARMS (Comprehensive Assessment of At-Risk Mental States) and its sub-assemblies : if the patient is at risk of psychosis, the test will classify this risk into one of the three following categories : group of trait and state risk factor, group of attenuated psychotic symptoms, group of BLIPS (Brief, Limited or Intermittent Psychotic Symptoms)
Results to tests concerning the peculiarities of cognitive functioning (neuropsychological assessment) assessed by Wechsler scale | Inclusion
  • Wechsler scale : neurocognitive assessment : Total intelligence quotient (between 60 and 140 approximately) Verbal comprehension index: 50 to 160 Perceptual reasoning index: 50 to 160 Working memory index: 50 to 160 Processing speed index: 50 to 160
Results to social functioning test: | Inclusion
  • Alterations in social functioning at SOFAS : Social and Occupational Functioning Assessment Scale : score theoretically between 0 and 100%. The lower the score, the worse the subject's functioning and therefore the higher the vulnerability.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LAVENNE, Principal Investigator — CHRU BREST
Locations (1):
- CHRU BREST Hôpital de Bohars, Bohars, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital (UH). Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Frith CD, Corcoran R. Exploring 'theory of mind' in people with schizophrenia. Psychol Med. 1996 May;26(3):521-30. doi: 10.1017/s0033291700035601. PMID 8733211
- [Background] Fusar-Poli P, Borgwardt S, Bechdolf A, Addington J, Riecher-Rossler A, Schultze-Lutter F, Keshavan M, Wood S, Ruhrmann S, Seidman LJ, Valmaggia L, Cannon T, Velthorst E, De Haan L, Cornblatt B, Bonoldi I, Birchwood M, McGlashan T, Carpenter W, McGorry P, Klosterkotter J, McGuire P, Yung A. The psychosis high-risk state: a comprehensive state-of-the-art review. JAMA Psychiatry. 2013 Jan;70(1):107-20. doi: 10.1001/jamapsychiatry.2013.269. PMID 23165428
- [Background] Thirioux B, Wehrmann M, Langbour N, Jaafari N, Berthoz A. Identifying Oneself with the Face of Someone Else Impairs the Egocentered Visuo-spatial Mechanisms: A New Double Mirror Paradigm to Study Self-other Distinction and Interaction. Front Psychol. 2016 Aug 25;7:1283. doi: 10.3389/fpsyg.2016.01283. eCollection 2016. PMID 27610095
- [Background] Keromnes G, Motillon T, Coulon N, Berthoz A, Du Boisgueheneuc F, Wehrmann M, Martin B, Thirioux B, Bonnot O, Ridereau R, Bellissant E, Drapier D, Levoyer D, Jaafari N, Tordjman S. Self-other recognition impairments in individuals with schizophrenia: a new experimental paradigm using a double mirror. NPJ Schizophr. 2018 Nov 28;4(1):24. doi: 10.1038/s41537-018-0065-5. PMID 30487540
- [Background] Keromnes G, Chokron S, Celume MP, Berthoz A, Botbol M, Canitano R, Du Boisgueheneuc F, Jaafari N, Lavenne-Collot N, Martin B, Motillon T, Thirioux B, Scandurra V, Wehrmann M, Ghanizadeh A, Tordjman S. Exploring Self-Consciousness From Self- and Other-Image Recognition in the Mirror: Concepts and Evaluation. Front Psychol. 2019 May 7;10:719. doi: 10.3389/fpsyg.2019.00719. eCollection 2019. PMID 31133909
- [Background] Uddin LQ, Davies MS, Scott AA, Zaidel E, Bookheimer SY, Iacoboni M, Dapretto M. Neural basis of self and other representation in autism: an FMRI study of self-face recognition. PLoS One. 2008;3(10):e3526. doi: 10.1371/journal.pone.0003526. Epub 2008 Oct 29. PMID 18958161
- [Background] Ionta S, Gassert R, Blanke O. Multi-sensory and sensorimotor foundation of bodily self-consciousness - an interdisciplinary approach. Front Psychol. 2011 Dec 23;2:383. doi: 10.3389/fpsyg.2011.00383. eCollection 2011. PMID 22207860
- [Background] Parnas J, Moller P, Kircher T, Thalbitzer J, Jansson L, Handest P, Zahavi D. EASE: Examination of Anomalous Self-Experience. Psychopathology. 2005 Sep-Oct;38(5):236-58. doi: 10.1159/000088441. Epub 2005 Sep 20. No abstract available. PMID 16179811